CLINICAL TRIAL: NCT02402998
Title: Eltrombopag as Second Line Therapy in Adult Patients With Primary Immune Thrombocytopenia (ESTIT Study) in an Attempt to Achieve Long-term Remission: a Single Arm Multicenter Phase II Clinical and Biological Study
Brief Title: Eltrombopag in Second Line Adult Primary Immune Thrombosytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP0815; 2015-001327-23 (EudraCT Number)
Record Dates: First submitted 2015-03-22; First posted 2015-03-31 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Primacy Immune Thrombocytopenia
Keywords: Primacy immune thrombocytopenia; Adults; Eltrombopag; Long-term remission
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag 50 mg/daily.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 50 mg/daily.

SUMMARY:
A clinical study to evaluate the efficacy of a drug called eltrombopag in adult patients affected of primary immune thrombocytopenia as first treatment to address the disease.

DETAILED DESCRIPTION:
This is a prospective, multicenter phase II trial designed to evaluate the activity of Eltrombopag second line treatment in adult patients with primary Immune Thrombocytopenia (ITP) not responsive or in relapse after a full first line steroids treatment (prednisone or dexamethasone) ± Intravenous Immune Globulin (IVIG).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary ITP;
2. Age ≥ 18 years;
3. Patients are in the new diagnosis or persistent phase of disease (i.e. within month 12 from diagnosis);
4. Patients not responsive or in relapse after a full course of steroid therapy (prednisone 1 mg/kg/d for at least 28 days or 3 cycles of dexamethasone 40 mg/day for consecutive 4 days, according to the GIMEMA ITP0207 trial) ± IVIG;
5. Patients have a platelet count < 10 x 109/L documented in a single blood cell count;
6. Patients have bleeding symptoms and a platelet count > 10 < 30 x 109/L documented in a single blood cell count;
7. Patients have no bleeding symptoms and a platelet count >10 < 30 x 109/L in at least 2 blood cell counts at 3 days interval in the week preceding the enrollment with the last count at the day of enrollment;
8. Patients have corticosteroids or IVIG dependence (the need for ongoing or repeated doses administration of corticosteroids or IVIG to maintain a platelet count ≥ 30 x 109/L and/or to avoid bleeding;
9. Written informed consent obtained from the subject;
10. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from time of enrollment until 6 months after the last dose of study treatment;
11. Female subjects of non-childbearing potential may be enrolled in the study; for this study population, non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause; OR
12. Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to start of Eltrombopag, has a negative pregnancy test within 14 days of first dose of Eltrombopag, and has agreed to continue adequate contraception during the entire treatment period and for 6 months after completion of the treatment.

Exclusion Criteria:

1. Diagnosis of secondary ITP. As far as patients with immune thrombocytopenia and antiphospholipid antibodies positivity, individuals without a previous thromboembolic event are excluded only if lupus anticoagulant (LAC) is associated with the presence of anticardiolipin (aCL) and aβ2-Glycoprotein I (aβ2GPI) antibodies;
2. Previous treatment with other anti-ITP second line therapies (i.e. Rituximab, Azathioprine, Cyclosporin-A or other); only patients with a previous full course of steroid (see inclusion criteria for definition) ± IVIG are admitted to the study;
3. Previous treatment with any TPO-R agonists;
4. Patients have life threatening bleeding complications;
5. Patients had deep venous thrombosis (DVT) or arterial thrombosis in the 3 months preceding the enrollment;
6. Patients are HIV, HCV, HBsAg positive;
7. Patients with hepatic impairment (i.e. mild, moderate or severe hepatic impairment (Child-Pugh score > 6);
8. Patients have a well established liver disease that represents a contraindication for the use of Eltrombopag;
9. Patients are unable to respect the 4-hour interval between Eltrombopag and other medications (e.g. antacids), calcium-rich foods (e.g. dairy products and calcium fortified juices), or supplements containing polyvalent cations such as iron, calcium, aluminium, magnesium, selenium, and zinc;
10. Patients are unable to stop medications that are known to cause a drug-drug interaction with Eltrombopag;
11. Subjects meeting any of the following criteria must not be enrolled in an Eltrombopag study:

    * Lactating female.
    * History of another malignancy. Exception: subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
    * Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the study procedures.
    * Hormone replacement therapy. Subjects must discontinue hormone replacement therapy prior to study enrollment due to the potential for inhibition of Cytochrome P450 (CYP) enzymes that metabolize estrogens and progestins.
    * Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment.
    * Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to Eltrombopag or excipients that contraindicate their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects who achieve long-term response (6 months sustained response) and able to taper down the dose. | After one year from study treatment.
  A patient will achieve this endpoint if at the end of the period of treatment he/she reaches to discontinue Eltrombopag and if, after discontinuation, has absence of bleeding and maintains a platelet count ≥ 30 x 109/L and at least a 2-fold increase from the baseline count in blood cell count performed in the 6 months of the period observation, during which no steroid, Eltrombopag, other anti TPO-R agonists and other anti-ITP medications are administered.

SECONDARY OUTCOMES:
Number of months of response from eltrombopag discontinuation to the last follow-up. | After one year from study treatment.
Number of months of complete response from eltrombopag discontinuation to the last follow-up. | After one year from study treatment.
Number of bleeding events. | After one year from study treatment.

OTHER OUTCOMES:
Modification of immunological parameters during treatment and their relationship with clinical outcomes. (Composite outcome) | At baseline, week 24, 36 and 52
  This study will be performed and completed in all patients enrolled into the study (responders and no-responders). The following biological markers will be evaluated from peripheral blood at baseline, week 24, 36 and 52:
  1. Cytokine serum levels;
  2. Lymphocyte subpopulations;
  3. Cytokine production by T cells ex vivo;
  4. Cytokine production by myeloid dendritic cells.
Analysis of the relationship between baseline TPO serum level and response to therapy. | After six months from treatment start.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Pr., Study Chair — Clinica Ematologica, DISM, Azienda Ospedaliera Universitaria S. M. Misericordia
Locations (14):
- Italy (14):
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - Azienda Ospedaliera "S.Gerardo", Monza
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - AO di Padova Università degli Studi Padova Dipartimento di Medicina Clinica Medica I - Medicina Interna CLOPD, Padua
  - Ospedale "Infermi", Rimini
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari Azienda Ospedaliero-Universitaria, Udine, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - Ospedale San Bortolo, Vicenza